CLINICAL TRIAL: NCT02080611
Title: Smart Textile Technology for Scoliosis: Aim 1
Brief Title: Smart Textile Technology for Scoliosis
Status: Withdrawn | Type: Observational
Why Stopped: Funding was not available from company
Sponsor: University of Minnesota (Other)
Collaborators: Moai Technologies (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1402M47947
Record Dates: First submitted 2014-02-28; First posted 2014-03-06 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Spinal Deformities; Scoliosis; Kyphosis
MeSH Terms: conditions — Scoliosis; Kyphosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesize that a garment-integrated sensing system will be able to detect with clinical accuracy the position of the spine. The investigator will evaluate this using healthy adult volunteers, who will don sensing garments and assume a series of spinal postures. Concurrent with garment sensing, the participant's spine position will be measured using a motion-capture system that uses reflective markers to detect positions of markers in 3D space.

The motion-capture system provides a gold-standard reference measure to which the sensing garments will be compared. Because the investigators are evaluating the accuracy of the sensing garment, it is only necessary that the investigator test the garments on participants with subtly different body shapes. Healthy adult volunteers provide an adequate input to the sensing signal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Under age 18 or over age 65
* Any medical condition that impairs movement or makes movement painful or difficult.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers will be used, recruited from the university community.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Body movement | Participants will be assessed during a 1-2 hour visit. Visits will be scheduled over a period of approximately one year.
  The movement and position of participants' spine will be recorded using a motion capture device and using a prototype sensing garment during the 1-2 hour lab test. (This is the only point at which investigators will interact with participants)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Dunn, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States